Dr Anushka Soni Botnar Research Centre, Windmill Road, Oxford, OX3 7LD Anushka.soni@ndorms.ox.ac.uk

T: 01865 227 374

| Study Code: | | Site ID Code: | | | _ | Participant identification number: |
|---|---|---|---|---|---|---|
| F | М | | 0 | Х | | PAIN |

## REMOTE CONSENT FORM

**Title:** Characterisation of **Pain** in patients with musculoskeletal disease: a prospective, Longitudinal, observational study with an **E**mbedded feasibility window of opportunity **S**leep **S**tudy (Pain-LESS)

## Name of Researcher:

Researcher to seek and record informed oral consent, after participant has had sufficient time to think about whether they want to take part.

Please check the boxes to record that the question has been asked by the researcher and that the participant has responded in the affirmative:

| 1) I confirm that I have read the information sheet dated03 May 23 (version7.1_) for this study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | |
|---|---|---|
| 2) I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | |
| 3) I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from University of Oxford, from regulatory authorities and from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | |
| 4) I understand that this is a research scan that is not useful for medical diagnosis, and that scans are not routinely looked at by a doctor. If a concern is raised about a possible abnormality on my scan, I will only be informed if a doctor thinks it is medically important such that the finding has clear implications for my current or future health. | | |
| | Yes | No |
| 5) I agree to donate blood samples. I consider these samples a gift to the University of Oxford and I understand I will not gain any direct personal or financial benefit from them. | | |
| | | No |
| 6a) I understand and agree that my samples will be used in research<br>aimed at understanding the genetic and molecular influences on disease<br>and that the results of these investigations are unlikely to have any<br>implications for me personally. | | |

Characterisation of **Pain** in patients with musculoskeletal disease: a prospective, **L**ongitudinal, observational study with an **E**mbedded feasibility window of opportunity **S**leep **S**tudy (Pain-LESS). Remote consent form, version 2.1, 03 May 2023. REC ref. 19/SC/0168. IRAS Project ID: 252762

| Ch) Lunderstand that the genetic analysis may identify recults which are | Yes | No |
|---|---|---|
| 6b) I understand that the genetic analysis may identify results which are found by chance (incidental findings) and/or medically actionable (judged to be important for my health and can be acted upon medically). I wish to be informed about such medically actionable genetic findings. | | |
| | Yes | No |
| 7) If invited, I agree to take part in some online games. | | |
| 8) If invited, I agree to be recorded whilst performing physio-type movements. | | No |
| 9) If invited, I agree to take part in an online sleep intervention with sleep monitoring. | | No |
| | Yes | No |
| 10a) I understand that if I am invited to participate in a focus group, an audio recording will be taken of the focus group in which I participate. | | |
| b) I agree to my statements in the focus group being quoted in the write up of this study. | | No |
| 11) I agree to take part in this study. | | |
| Additional: | | |
| 12) I agree to be contacted about ethically approved research studies for | Yes | No |
| which I may be suitable. I understand that agreeing to be contacted does not oblige me to participate in any further studies. | | |
| 40) Leaves for my approximated consider to be used in fature as | | No |
| 13) I agree for my anonymised samples to be used in future research,<br>here or abroad, which has ethics approval. I understand this research may<br>involve commercial organisations. | | |
| Name of Participant | | |

\*1 for participant (e.g. emailed securely to participant); 1 for researcher site file (original); 1 (to be kept in medical notes (if participant is a patient).

Date

Characterisation of **Pain** in patients with musculoskeletal disease: a prospective, **L**ongitudinal, observational study with an **E**mbedded feasibility window of opportunity **S**leep **S**tudy (Pain-LESS). Remote consent form, version 2.1, 03 May 2023. REC ref. 19/SC/0168. IRAS Project ID: 252762

Name of Researcher taking consent

Signature